CLINICAL TRIAL: NCT02843256
Title: Changes in CO2-13/CO2-12 Delta Value in Exhaled Breath to Examine Changes in Metabolism in Patients Being Fed Intravenous Nutrition
Brief Title: Using Exhaled Air to Determine Changes in Nutritional Status of Patients on Intravenous Nutrition
Acronym: UEAIVN
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Isomark, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-0354
Record Dates: First submitted 2016-06-06; First posted 2016-07-25 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Malnourished; Fasting
MeSH Terms: conditions — Obesity; Malnutrition; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving intravenous nutrition: Patients will blow into a bag that will capture 500 mL of their exhaled air daily for 7 days or the length of the parenteral nutrition, whichever is shorter. The Isomark Canary will analyze the air to generate a breath delta value.
  Interventions: Device: Isomark Canary

INTERVENTIONS:
Device: Isomark Canary — The Isomark Canary will analyze the exhaled air and generate a breath delta value.

SUMMARY:
Carbon-12 and carbon-13 are naturally-occurring isotopes that are found in exhaled breath. Investigators have proved that the 13CO2/12CO2 breath delta value (BDV) changes in subjects who were in negative energy balance then fed a positive energy balance meal. Measuring one liter of exhaled breath daily may be a more convenient way to measure negative or positive energy balance in patients receiving intravenous nutrition.

DETAILED DESCRIPTION:
This is a prospective, pilot study to determine if there is change in the 12C/13C BDV between days 0-7 in patients who receive parenteral nutrition. Investigators will recruit subjects from inpatient units at the University of Wisconsin Hospital and Clinics whose primary team consult the Nutrition Support Team to institute parenteral nutrition for clinical reasons. Subjects with clinical indications for parenteral nutrition are moderately to severely malnourished due to little to no nutrition by other means (oral nutrition or nutrition per tube) for a period of time (0-10 days based on state of nourishment prior to admission).

Investigators will record baseline nutritional status from the medical record notes (dietitian, Nutrition Support Team, etc.), as well as medication, demographic information and medical history. Investigators will take a baseline exhaled CO2 measurement and then a daily measurement at approximately the same time daily (+/- an hour).

The daily exhaled 12C/13C breath delta value will be matched with the subjects' daily caloric intake from parenteral nutrition (and oral nutrition and nutrition per tube, if applicable). The breath delta value, the caloric intake, plus the subjects' degree of malnourishment will be parameters with which to build further research. Investigators hypothesize that the breath delta value will increase from baseline and then stabilize after the patient reaches goal energy needs as defined by the Nutrition Support Team.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Anticipated start of parenteral nutrition
* Expected duration of stay at least 5 days from enrollment
* Subject speaks English
* Subjects with inability to take adequate oral nutrition who are developing or have developed malnutrition who require parenteral nutrition

Exclusion Criteria:

* Subjects unable to coordinate well enough to give a 1 liter breath sample
* Subjects receiving parenteral nutrition prior to admission
* Subjects who are pregnant
* Subjects who are prisoners
* Subjects who are pharmacologically sedated or with altered consciousness
* Subjects who are mechanically ventilated
* Subjects admitted for bone marrow or stem cell transplants
* Known participation in another interventional research study within 30 days prior to enrollment (note: to be eligible, any interventional treatment must have ended at least 30 days ago)
* Subjects with disease states or clinical conditions that do not make them study candidates, per the primary investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age 18 or order) with clinical indications for parenteral nutrition who are moderately to severely malnourished due to little to no nutrition by other means (oral nutrition or nutrition per tube) for a period of time (0-10 days based on state of nourishment prior to admission).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Variation in Breath Delta Value | baseline to day 7
  Investigators will test if the breath delta value (kJ) increases in subjects from baseline (pre-parenteral nutrition) to the subject's goal calculated rate. The time frame tested for each subject will be from baseline to 7 days or the length of parenteral nutrition (whichever is shorter.) Investigators will recruit 20 patients, and this may take 6 months to accomplish. This is a pilot investigation.

SECONDARY OUTCOMES:
Variation in Breath Delta Value from day 0 to day 1 of parenteral nutrition | day 0 to day 1
  Investigators hypothesize that the variation in breath delta value (kJ) will show the most dramatic change in subjects receiving parenteral nutrition from baseline to day 1 of parenteral nutrition.
Subjects and Variation in Breath Delta Value | baseline to day 7
  Investigators hypothesize that the variation in breath delta value (kJ) will show the most variation from baseline to day 7 in subjects who are the most malnourished (that is, the subjects who have lost the most weight prior to starting parenteral nutrition)
Variation in Breath Delta Value when Parenteral Nutrition is interrupted | baseline to day 7
  Investigators hypothesize that there will be a variation in breath delta value (kJ) if parenteral nutrition is interrupted (for clinical purposes, that is, due to a central line infection or other clinical reason.)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Kudsk, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided